CLINICAL TRIAL: NCT06266767
Title: Programmed Intermittent Epidural Bolus (PIEB) Techniques for Labour Analgesia; Finding the Optimum Combination
Brief Title: Programmed Intermittent Epidural Bolus (PIEB) Techniques for Labour Analgesia
Acronym: PIEB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Health Services Research
Other Study IDs: MRC-01-18-157
Record Dates: First submitted 2023-11-19; First posted 2024-02-20 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Labor Pain; Obstetric Pain; Analgesia
Keywords: Obstetrics; Analgesia; Epidural; Patient-Controlled; Opioid
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Levobupivacaine; Fentanyl

STUDY DESIGN:
Intervention Model Description: We aim to use a pragmatic sequential optimization method as described by Sveticic et al. 2003. For the first round of recruitment, the research team will randomize women into 8 different groups of PIEB/PCEA regimens with six (n=6) women per group and set up the epidural pump for the maintenance of labor analgesia. This first round of recruitment will be called Complex #1. The PCEA bolus volume and lockout interval will stay the same for all groups.
  There will be 8 combinations of PIEB/PCEA using an epidural mixture of 0.1% levobupivacaine + 2mcg/ml Fentanyl (n=48). We will exclude the 2 worst performing groups (as assessed by our composite primary outcome). Using sequential optimization, 2 new groups with different combinations of PIEB volume / interval will be added to the remaining 6 groups. Complex 2 therefore will consist of 8 groups of 48 patients (n=6 per group). We anticipate 3 to 4 rounds of recruitment until our statistician determines the 2 best performing groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This is a randomized double-blinded design. Patients and their attending physicians / clinical anaesthetists / data collection study member / midwives / nurses will be blinded to patient group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Group 1 (Experimental): PIEB bolus vol (ml) : 8 PIEB time interval (min) : 60 PCEA bolus vol (ml) : 5 PCEA lockout time interval (min) : 20
  Interventions: Drug: Levobupivacaine and Fentanyl
- Group 2 (Experimental): PIEB bolus vol (ml) : 8 PIEB time interval (min) : 45 PCEA bolus vol (ml) : 5 PCEA lockout time interval (min) : 20
  Interventions: Drug: Levobupivacaine and Fentanyl
- Group 3 (Experimental): PIEB bolus vol (ml) : 10 PIEB time interval (min) : 30 PCEA bolus vol (ml) : 5 PCEA lockout time interval (min) : 20
  Interventions: Drug: Levobupivacaine and Fentanyl
- Group 4 (Experimental): PIEB bolus vol (ml) : 10 PIEB time interval (min) : 45 PCEA bolus vol (ml) : 5 PCEA lockout time interval (min) : 20
  Interventions: Drug: Levobupivacaine and Fentanyl
- Group 5 (Experimental): PIEB bolus vol (ml) : 10 PIEB time interval (min) : 60 PCEA bolus vol (ml) : 5 PCEA lockout time interval (min) : 20
  Interventions: Drug: Levobupivacaine and Fentanyl
- Group 6 (Experimental): PIEB bolus vol (ml) : 10 PIEB time interval (min) : 75 PCEA bolus vol (ml) : 5 PCEA lockout time interval (min) : 20
  Interventions: Drug: Levobupivacaine and Fentanyl
- Group 7 (Experimental): PIEB bolus vol (ml) : 12 PIEB time interval (min) : 60 PCEA bolus vol (ml) : 5 PCEA lockout time interval (min) : 20
  Interventions: Drug: Levobupivacaine and Fentanyl
- Group 8 (Experimental): PIEB bolus vol (ml) : 12 PIEB time interval (min) : 45 PCEA bolus vol (ml) : 5 PCEA lockout time interval (min) : 20
  Interventions: Drug: Levobupivacaine and Fentanyl

INTERVENTIONS:
Drug: Levobupivacaine and Fentanyl — Programmed Intermittent Epidural Bolus

SUMMARY:
Epidural Analgesia remains the most effective form of pain relief in labour. After initiating epidural analgesia, there are many epidural drug regimens that can be employed to maintain analgesia for the duration of labour using an epidural catheter. Due to recent advances in medical technology, new epidural pumps, which allow both patient controlled epidural analgesia boluses (PCEA, a common standard of care in many hospitals) and programmed intermittent epidural boluses (PIEB, automatic boluses given in addition to the PCEA bolus), are now available. In this randomized double-blind trial, we aim to evaluate the effects of different combinations of PIEB (epidural bolus volume) and PIEB (bolus volume and time interval) on labour patient-controlled epidural analgesia (PCEA) usage. In theory, the more effective the PIEB combination (the ideal drug volume and ideal time interval), the less PCEA boluses (extra epidural drug) will be used as well as less clinician boluses and less lower limb weakness (motor block) as assessed by the Bromage Score.

DETAILED DESCRIPTION:
Many women experience severe pain during labour. There are many forms of pain relief methods available to women in developed countries. Labour epidural analgesia remains the most effective form of pain relief. It is also the least depressive to the central nervous system of the mother and the baby. After initiating epidural analgesia, there are many regimens that can be employed to maintain analgesia for the duration of labour.

Traditionally, epidural analgesia (using low dose mixtures of local anaesthetic and opioid) has been administered by nurse or midwife-controlled manual boluses or as continuous infusion via a dedicated epidural pump (once the epidural catheter has been placed by an anaesthetist). Although these regimens provide an effective form of labour analgesia, patient satisfaction is not always achieved because of the associated lower limb motor block (leg weakness) and the increased risk of requiring instrumental delivery such as a forceps delivery. Due to recent advances in medical technology, new epidural pumps, which allow patient controlled epidural analgesia (PCEA) boluses and programmed intermittent epidural (PIEB) boluses, are now available.

Bolus injection through an epidural catheter may result in better distribution of anaesthetic solution in the epidural space when compared with continuous infusion of the same low dose local anaesthetic / opioid mixture. Capogna et al carried out a randomized double-blind study to compare the effects of a programmed intermittent epidural bolus (PIEB) regimen with a continuous epidural infusion (CEI). Motor block was reported in 37% in the CEI group and in only 2.7% in the PIEB group (P < 0.001). The incidence of instrumental delivery was 20% for the CEI group and 7% for the PIEB group (P = 0.03). The total local anaesthetic consumption, number of patients requiring additional PCEA boluses, and mean number of PCEA boluses per patient were also found to be lower in the PIEB group (P < 0.001). There were no differences in pain scores and duration of labour analgesia. (Capogna et al, 2011) Another randomized controlled study published by Wong et al compared total local anaesthetic (bupivacaine was used in this study) consumption, need for supplemental epidural analgesia, quality of analgesia, and patient satisfaction in women who received programmed intermittent epidural boluses (PIEB) compared with continuous epidural infusion (CEI) for maintenance of labour epidural analgesia. The median total bupivacaine dose per hour of analgesia was significantly less in the PIEB (n = 63) (10.5 mg/h; 95% confidence interval, 9.5-11.8 mg/h) when compared with the CEI group (n = 63) (12.3 mg/h; 95% confidence interval, 10.5-14.0 mg/h) (P < 0.01). Patient satisfaction scores were also higher in the PIEB group. The authors concluded that PIEB combined with patient controlled epidural analgesia (PCEA) provided similar analgesia, but with a smaller bupivacaine dose and better patient satisfaction compared with CEI with PCEA for maintenance of epidural labour analgesia. (Wong et al, 2006) Wong et al carried out another study to evaluate bupivacaine consumption and other analgesic outcomes when the programmed intermittent bolus time interval and volume were manipulated during the maintenance of epidural labour analgesia. They found that extending the programmed intermittent bolus interval and volume from 15 minutes to 60 minutes, and 2.5 mL to 10 mL, respectively, decreased bupivacaine consumption without decreasing patient comfort or satisfaction. (Wong et al, 2011) In our study, we aim to compare the effects of different combinations of PIEB bolus volume and PIEB time interval on the number of PCEA demands / clinician boluses, pain score, local anaesthetic consumption and patient satisfaction in order to find the optimal PIEB volume and PIEB time interval for labour pain relief when used together with a fixed (pre-determined) PCEA regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 yrs
* In active labour
* ASA 2 patients (pregnant patients are considered to be ASA 2)
* Singleton pregnancy
* > 37 weeks gestation
* Booking BMI 18 to 35

Exclusion Criteria:

* BMI < 18
* BMI > 35
* Systemic opioids within the previous 6 hours
* Presence of a fetal anomaly
* Pre-eclampsia
* Bleeding disorders (including coagulation disorders)
* Recent spinal surgery
* Spinal injury
* Elevated intracranial pressure (ICP)
* Neuraxial disorders of any description
* Signs of local or systemic infection
* Patient refusal for neuraxial analgesia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — parturient 37+ weeks
Enrollment: 136 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
The volume of local anaesthetic mixture for breakthrough pain (PCEA + clinician bolus) + the Bromage Score | From the siting of the epidural block to the delivery of the fetus (maximum 24 hrs)
  The (composite) primary outcome will identify the 2 best performing groups

SECONDARY OUTCOMES:
Pain score | From the siting of the epidural block to the delivery of the fetus (maximum 24 hrs)
  Numeric Rating Scale (NRS). Patient self-reported pain scale. 0 (No Pain) to 10 (Worst possible pain)
Total local anesthetic consumption | From the siting of the epidural block to the delivery of the fetus (maximum 24 hrs)
  Initial Epidural Bolus + Total volume PIEB + Total volume PCEA + Clinician bolus volume
Need for supplementary epidural analgesia | From the siting of the epidural block to the delivery of the fetus (maximum 24 hrs)
  Total volume PCEA + Total volume clinician Bolus
Bromage score (lower limb weakness score) | From the siting of the epidural block to the delivery of the fetus (maximum 24 hrs)
  Bromage Score -1: Free movement of legs and feet, 2: Just able to flex knees, able to move feet, 3: Unable to flex knees, able to move feet, 4 :Unable to move legs or feet
Type of delivery | From the siting of the epidural block to the delivery of the fetus (maximum 24 hrs)
  Normal vaginal delivery, cesarean delivery, forceps and vacuum delivery
Sensory block | From the siting of the epidural block for 3 hours
  Assessed with cold spray (ethyl chloride)
Fetal Outcome | At the time of birth and 5 minutes after delivery
  Umbilical cord blood gases + Apgar scores

CONTACTS AND LOCATIONS:
Overall Officials: Roshan Fernando, MD, Principal Investigator — Hamad Medical Corporation, Qatar; Fatima Khatoon, DESAIC, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation (HMC), Doha, Baladīyat ad Dawḩah, Qatar